CLINICAL TRIAL: NCT06409208
Title: Postnatal Care and Services Utilization in Nepal: Use of mHealth Intervention in Improving Utilization of Postpartum Care
Brief Title: Use of mHealth Intervention in Improving Utilization of Postpartum Care
Acronym: mHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dhulikhel Hospital (Other)
Responsible Party: Principal Investigator, Subasna Shrestha, Associate Professor, Dhulikhel Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHRC 36/2024
Record Dates: First submitted 2024-05-04; First posted 2024-05-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Postnatal Care
Keywords: mHealth Intervention
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, mHealth intervention (video and reminder SMSs) (Experimental): Intervention group of postnatal mothers will get mHealth intervention package which will include video on postnatal care and 13 reminder short text messages (SMS) which will be delivered to women different days of postnatal period. Reminder SMSs will be focused on Postnatal visits, post partum family planning and exclusive breast feeding practice.
  Interventions: Behavioral: mHealth intervention (video and reminder SMSs)
- Control arm (No Intervention): Routine antenatal and postnatal care

INTERVENTIONS:
Behavioral: mHealth intervention (video and reminder SMSs) — intervention includes educational video related to postnatal care and reminder SMSs related to postnatal visits, family planning adoption and exclusive breast feeding practice.
  Arms: Intervention, mHealth intervention (video and reminder SMSs)

SUMMARY:
Despite implementation of many activities related to maternal health, maternal mortality ratio is still unacceptably high in Nepal, 239/100,000 in live births. Most maternal deaths occur within 48 hours of delivery (42.7%) and then in the late postpartum period (from 48 hours after birth to up to six weeks after childbirth) (29.5%), postpartum hemorrhage predominate as the most important cause of maternal deaths (23%), with hypertensive disorder (eclampsia/pre-eclampsia) at 14 percent.

Postnatal care service is important for prevention of postnatal complications and to reduce maternal mortality. However, postnatal care service is rare in Nepal. And where it is available quality is poor. Forty-two (42%) percent of women did not receive any postnatal check in Nepal. Lack of awareness of importance to postnatal care, distance of health facility, unsuccessful endorsement of postnatal care by Government and cultural practice of Nepal are major causes of failure to attend postnatal care and visit in Nepal. Mhealth intervention would be the best option to address these constrains to attain or improve postnatal visits according to national protocol.

A qualitative and quantitative study will be conducted. Qualitative study will be conducted as a formative study to explore enabling and barriers to attend postnatal care visit. A focused group discussion will be done among postnatal mothers attending immunization clinic and gynae out patient department (OPD) of Dhulikhel hospital. A COM-B model of behavior change will be applied to identify enablers and barriers among women by conducting focus group discussions. Semi structured topic guide will be developed using sources of behaviors, capability, opportunity and motivation and its sub categories. Intervention package will be designed based on evidence that will support the use of behavioral theory for effective outcomes. Thematic Analysis of barriers and enablers to increase uptake of postnatal care (post natal visits, family planning and exclusive breast feeding) will be done by using same model.

A quantitative study will be conducted among antenatal mothers attending ANC clinic of tertiary care hospital. A randomized control trial method will be used for the study. Total of 300 third trimester antenatal women will be enrolled for the study. Intervention group will received intervention package which includes, health care video related to postnatal care, care of newborn, danger signs etc. This video will be shown to women during their antenatal period for the first time and then video will be downloaded to their respective mobile phone and will be motivated to watched them later at least for minimum of 3 times. Educational reminder messages will be sent to women around 13 times different periods of postpartum days. These SMSs will be mainly focused on reminder for postnatal care visits, use of postpartum family planning methods and importance of exclusive breast feeding practices. Control group will receive a standard care. At the end, health related outcomes will be measured in both groups as numbers of postnatal visit attended, use of postnatal family planning methods, exclusive breast feeding and seeking care for danger signs of mother and newborns by both groups will be evaluated. Implementation outcomes of mHealth intervention strategy will be evaluated using PROCTORs framework.

DETAILED DESCRIPTION:
A qualitative and quantitative study will be conducted. Qualitative study will be conducted as a formative study to explore enabling and barriers to attend postnatal care visit. A focused group discussion (FGD) will be done among postnatal mothers attending immunization clinic and gynecologic OPD of Dhulikhel Hospital. About 4 sessions of FGDs will be conducted. However, it will be based on data saturation. Once the data saturation is confirmed extra one more FGD will be conducted for new information.

A COM-B model components of behavior change wheel will be applied to identify enablers and barriers among women by conducting focus group discussions.1 Semi structured topic guide will be developed using sources of behaviors e.g. capability, opportunity and motivation and its sub components. Capability component comprises psychological and physical capabilities. Capability refers to an individual's psychological (mental skills and knowledge) and physical ability (bodily functions) to engage in a behavior. Opportunity component comprises physical and social sub components. Physical opportunity refers to the environment where the behavior takes place and social opportunity deals with social values, culture and social support. Motivation involves reflective and automatic motivation. Reflective motivation involves evaluation and plans and automatic motivation involves emotions and impulses.1 Based on these components topic guides for FGDs will be developed to explore barriers and enablers of postnatal care and visits.

Intervention package will be designed based on evidence that will support the use of behavioral theory for effective outcomes. After developing intervention package, before implementation the intervention package will be validated by experts' team and data safety and management board (DSMB) team. A half day workshop will be conducted. The expert team will include, HOD of gynecology and obstetrics department, obstetric consultant, Nurse manager and in-charge of Antenatal care clinic and postnatal ward and midwives of antenatal clinic. Thematic Analysis of barriers and enablers to increase uptake of postnatal care (post natal visits, family planning and exclusive breast feeding) will be done by using same model.

A quantitative study will be conducted among antenatal mothers attending ANC clinic of tertiary care hospital. A randomized control trial method will be used for the study. About 300 eligible pregnant women of third trimester visiting antenatal OPD of Dhulikhel Hospital will be enrolled for the study after consenting to participate. These women will be divided in to two groups as intervention group and control group.

The participants in each group will be randomly assigned to intervention and control group in 1:1 ratio.

Research assistant and researcher will explain each consenting woman and take them to a quite and private room to conduct a 30 minutes face to face interview to obtain the baseline information (demographic, obstetric information and postnatal care knowledge assessment) from the study participants from both groups with Postnatal care knowledge assessment will be done by Red cap app using tablets device.

Intervention group will receive intervention package which includes, health care video related to postnatal care, care of newborn, danger signs etc. This video will be shown to women during their antenatal period for the first time and then video will be downloaded to their respective mobile phone and will be motivated to watched them later at least for minimum of 3 times. Women will be called to watch video on 15 days of post partum for confirmation.

The second intervention package will include educational and reminder messages to women in different period of times. Educational reminder messages will be sent to women around 13 times different periods of postpartum days. These SMSs will be mainly focused on reminder for postnatal care visits, use of postpartum family planning methods and importance of exclusive breast feeding practices. Control group will receive a standard care. The first postnatal reminder SMS will be sent to women once she is identified as she had given birth, on the day of delivery. Second SMS will be delivered to women on third day of postpartum, consecutive SMS will be sent on 7th day, 10th day, 14th day, 40th day and 42nd days of postpartum respectively. This reminder SMSs are planned according to WHO recommendation of postpartum visit.2 (SMS will be sent on 2days prior to recommended visit and early morning of very right day of the visit) The third reminder and educational SMS will be related to exclusive breast feeding. This SMS will be delivered to women on day of delivery then, 15th day of postpartum and 30th day of postpartum. Next message related to family planning uptake will be sent to woman during antenatal period followed by 15th day and 30th day of postpartum to encourage to use postpartum family planning methods.

Follow up and end assessment,

At the end, health related outcomes will be measured in both groups as numbers of postnatal visit attended, use of postnatal family planning methods, exclusive breast feeding and seeking care for danger signs of mother and newborns by both groups will be evaluated. Implementation outcomes, acceptability, adoption, appropriateness, costs, feasibility, fidelity, penetration and sustainability of mHealth intervention strategy will be evaluated using PROCTORs framework.3

Additionally, feasibility of use of mHealth intervention among postnatal mothers will be measured by the system usability scale (SUS).4 The System Usability Scale (SUS) is a reliable and widely-used tool for global assessments of systems usability that contains 10 five-point Likert type questions.5

Data Analysis

Descriptive analysis. The descriptive statistics for baseline characteristics comparing intervention and control groups will be presented as frequencies (percent) for categorical variables and means (standard deviations) for continuous variables Comparison of characteristics of intervention and control group. We will be conducted an independent sample t-test to compare the continuous demographic and obstetric data, including age, income, family size, and first age at menarche, a gestational week at enrollment, and number of ANC visits between the intervention and comparison groups. A chi-square test will be used to compare group differences in categorical variables, including level of education, ethnicity, religion, occupation, frequency of TV and radio views, pregnancy intention, menstrual cycle, gravida, and parity.

Logistic regression model will be used for binary outcome variables, i.e., attendance of all four postnatal care visits (yes, no), use of family planning methods after birth (Yes, No), exclusive breast feeding practice (yes, no) by women in each group. Negative binomial regression model will be applied for postnatal visit counts by women. STATA software version 14.will be used for data analysis.

In addition, the investigators will analyze implementation outcomes, acceptability, appropriateness, adoption, fidelity, costs, penetration and sustainability by adapting PROCTORs framework which will be measured by qualitative approach (in-depth interview with participants) and quantitative approach (records of postnatal care clinics) with appropriate 95% confidence intervals.

Definition of Implementation outcomes

Acceptability- The perception that a mHealth intervention is agreeable and satisfactory or palatable to postnatal mothers.

Adoption- The Intention of postnatal mother to use mHealth intervention Appropriateness- The perceived fit or value of mHealth intervention to postnatal mothers Feasibility- The extent to which mHealth intervention can be used or carried out by postnatal mothers within a setting (ANC clinic and their homes).

Fidelity- The degree to which mHealth intervention is implemented as prescribed in the original protocol.

Costs- Cost for mHealth development, validation and implementation. Cost might include, app development, video development, development of SMS and delivery of it.

Penetration- Integration of mHealth intervention in to regular service setting Sustainability- The extent to which a mHealth intervention becomes part of normal practice.

Implementation outcome measurement

* Acceptability- The perception that a mHealth intervention is agreeable and satisfactory will be measured through in-depth interview among postnatal women participated in intervention group. Question- How acceptable do you feel using mHealth package? Time duration 6 month
* Adoption- The Intention of postnatal mother to use mHealth intervention. It will be measure by Proportion of women intended to use mHealth intervention / Total number of PNC mothers who will receive mHealth Intervention.
* Appropriateness- The perceived fit or value of mHealth intervention to postnatal mothers will be measured by in-depth interview. Question- How do you find mHealth intervention appropriate to understand?
* Feasibility- The extent to which mHealth intervention can be used or carried out by postnatal mothers within a setting (ANC clinic and their homes). It will be measured by % of PNC mothers using mobile apps in ease/ Total number of PNC mothers in intervention group. The System Usability Scale (SUS) will be used.5
* Fidelity- The degree to which mHealth intervention is implemented as prescribed in the original protocol. This will be measured by % of mothers watched video and received SMSs as per protocol/ total number of postnatal mother enrolled for intervention group in the study.
* Costs- cost for mHealth development, validation and implementation. Cost might include, app development, video development, development of SMS and delivery of it.
* Penetration- integration of mHealth intervention in to regular service setting will be measured by % of postnatal mothers will receive mHealth intervention / total number of postnatal women discharge from the hospital.
* Sustainability- The extent to which a mHealth intervention will be maintained or becomes part of normal practice. It will be measured by % of PNC mothers received mHealth intervention in 1year period/ total number of postnatal mothers delivered at Dhulikhel Hospital

Clinical outcomes

1. Postnatal visits attended-
2. Use Postpartum family planning methods
3. Exclusive breast feeding practice
4. Knowledge on postnatal care- pre and post knowledge assessment will be done

ELIGIBILITY:
Inclusion Criteria:

* - Women age 19 years and above
* III trimester pregnant lady
* Mobile phone user and able to read and understand Nepali language
* Literate and can operate mobile phone (can check text message and read)

Exclusion Criteria:

* - Women only come for child birth service at DH without attending ANC clinic of DH.
* Women with very sick newborn and neonatal death
* Women who has to stay hospital for longer period of time (more than 14 days)
* Women with complication during labour and delivery eg. Uterine rupture,
* Not able to come for delivery at Dhulikhel Hospital.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
uptake of postnatal visits | 6 weeks
  proportion of participants attended postnatal care clinic as per world health organization (WHO) recommendation (24 hours of child birth, 3days , 7-14 days and on 42days of post partum)
postpartum family planning adoption | 3 months
  proportion of participants used modern family planning methods
exclusive breast feeding practice | 3 months
  proportion participants exclusively breastfeeding her newborns

SECONDARY OUTCOMES:
Acceptability of mHealth Intervention | 3 months
  The perception that a mHealth intervention is agreeable and satisfactory will be measured through in-depth interview among postnatal women participated in intervention group. Question- How acceptable do you feel using mHealth package?
Adoption of mHealth Intervention | 3 months
  The Intention of postnatal mother to use mhealth intervention. It will be measure by Proportion of women intended to use mHealth intervention
Appropriateness of mHealth Intervention | 3 months
  The perceived fit or value of mHealth intervention to postnatal mothers will be measured by in-depth interview. Question- How do you find mHealth intervention appropriate to understand?
Feasibility of mHealth Intervention | 3 months
  The extent to which mHealth intervention can be used or carried out by postnatal mothers within a setting (ANC clinic and their homes). It will be measured by % of PNC mothers using mobile apps in ease
Penetration of mHealth Intervention | 3 months
  integration of mHealth intervention in to regular service setting will be measured by % of postnatal mothers will receive mHealth intervention
Sustainability of mHealth Intervention | 3 months
  The extent to which a mHealth intervention will be maintained or becomes part of normal practice. It will be measured by %of PNC mothers received mHealth intervention in 1year period

OTHER OUTCOMES:
knowledge on postnatal care | 3 months
  proportion of participants scoring 80% of knowledge on postnatal care

CONTACTS AND LOCATIONS:
Locations (1):
- Dhulikhel Hospital, Kathamandu University Hospital, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
all collected information

REFERENCES:
- [Background] Dhakal S, Chapman GN, Simkhada PP, van Teijlingen ER, Stephens J, Raja AE. Utilisation of postnatal care among rural women in Nepal. BMC Pregnancy Childbirth. 2007 Sep 3;7:19. doi: 10.1186/1471-2393-7-19. PMID 17767710
- [Background] Sharma S, van Teijlingen E, Hundley V, Angell C, Simkhada P. Dirty and 40 days in the wilderness: Eliciting childbirth and postnatal cultural practices and beliefs in Nepal. BMC Pregnancy Childbirth. 2016 Jul 5;16(1):147. doi: 10.1186/s12884-016-0938-4. PMID 27381177
- [Background] Lama TP, Munos MK, Katz J, Khatry SK, LeClerq SC, Mullany LC. Assessment of facility and health worker readiness to provide quality antenatal, intrapartum and postpartum care in rural Southern Nepal. BMC Health Serv Res. 2020 Jan 6;20(1):16. doi: 10.1186/s12913-019-4871-x. PMID 31906938
- [Background] Adanikin AI, Awoleke JO, Adeyiolu A. Role of reminder by text message in enhancing postnatal clinic attendance. Int J Gynaecol Obstet. 2014 Aug;126(2):179-80. doi: 10.1016/j.ijgo.2014.02.009. Epub 2014 Apr 2. No abstract available. PMID 24794692
- [Background] Olajubu AO, Fajemilehin BR, Olajubu TO, Afolabi BS. Effectiveness of a mobile health intervention on uptake of recommended postnatal care services in Nigeria. PLoS One. 2020 Sep 14;15(9):e0238911. doi: 10.1371/journal.pone.0238911. eCollection 2020. PMID 32925971
- [Background] Unger JA, Ronen K, Perrier T, DeRenzi B, Slyker J, Drake AL, Mogaka D, Kinuthia J, John-Stewart G. Short message service communication improves exclusive breastfeeding and early postpartum contraception in a low- to middle-income country setting: a randomised trial. BJOG. 2018 Nov;125(12):1620-1629. doi: 10.1111/1471-0528.15337. Epub 2018 Aug 28. PMID 29924912
- [Background] Beraki GG, Tesfamariam EH, Gebremichael A, Yohannes B, Haile K, Tewelde S, Goitom S. Knowledge on postnatal care among postpartum mothers during discharge in maternity hospitals in Asmara: a cross-sectional study. BMC Pregnancy Childbirth. 2020 Jan 6;20(1):17. doi: 10.1186/s12884-019-2694-8. PMID 31906883
- [Background] Chaudhary K, Nepal J, Shrestha K, Karmacharya M, Khadka D, Shrestha A, Shakya PR, Rawal S, Shrestha A. Effect of a social media-based health education program on postnatal care (PNC) knowledge among pregnant women using smartphones in Dhulikhel hospital: A randomized controlled trial. PLoS One. 2023 Jan 20;18(1):e0280622. doi: 10.1371/journal.pone.0280622. eCollection 2023. PMID 36662821
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] martins et al. European Portuguese Validation of the System Usability Scale (SUS) https://linkinghub.elsevier.com/retrieve/pii/S1877050915031191
- [Background] WHO recommendations on maternal and newborn care for a positive postnatal experience [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK579657/ PMID 35467813
- [Result] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- See also: World Health Organization. Trends in maternal mortality 2000 to 2020: estimates by WHO, UNICEF, UNFPA, World Bank Group and UNDESA/Population Division [Internet]. Trends in maternal mortality 2000 to 2020. 2023 — https://www.who.int/publications-detail-redirect/9789240068759
- See also: MOH/Nepal M of H, ERA/Nepal N, ICF. Nepal Demographic and Health Survey 2016. 2017 Nov 1 — https://dhsprogram.com/publications/publication-fr336-dhs-final-reports.cfm